CLINICAL TRIAL: NCT03658161
Title: Communicating About Sexual Concerns and Dysfunction Effectively (CASCADE) Program
Acronym: CASCADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00071979
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CASCADE (Experimental): Oncology providers will receive the CASCADE coaching intervention.
  Interventions: Behavioral: Communicating About Sexual Concerns and Dysfunction Effectively

INTERVENTIONS:
Behavioral: Communicating About Sexual Concerns and Dysfunction Effectively — The coaching intervention will include two parts: 1) initial coaching session, and 2) follow-up appointment to check in on use of the intervention strategies.
  Other Names: CASCADE

SUMMARY:
Patients with cancer suffer many devastating side effects; one that is understudied but vital to quality of life is the effect of cancer and its treatments on patients' sexual functioning and satisfaction. The long-term goal of this work is to improve the care of patients with cancer who are experiencing difficulties with sexual function and satisfaction. As a necessary first step, providers must be skilled in eliciting patients' concerns about sexual health and addressing them appropriately. However, prior studies have found that (1) oncology providers are reluctant to discuss sexual issues with their patients, (2) patients report that needed conversations about their sexual concerns do not occur, and (3) patients want to discuss sexual health with their provider. Thus, the goal of the present study is to develop and test a brief intervention to improve oncology provider's skills in addressing patients' concerns regarding sexual function-the Communicating about Sexual Concerns and Dysfunction Effectively (CASCADE) Program.

To aid in development of the intervention, focus groups will be held and target 9 distinct populations of cancer survivors: 1) Breast; 2) Gynecologic; 3) Prostate; 4) males with gastrointestinal malignancies; 5) females with gastrointestinal malignancies; 6) males with brain tumors; 7) females with brain tumors; 8) LGBTQ individuals who identify as male; 9) LGBTQ individuals who identify as female. Maximum accrual for this phase will be 90 patients for 9 focus groups, or a maximum of 10 patients per group. Groups will last approximately 75 minutes and be audio recorded. Participants will also complete self-report measures which as about their sexual functioning, emotional wellbeing, physical functioning and utilization of services offered through the Duke Cancer Institute.

The intervention will then be pilot tested with up to 10 providers to assess feasibility and acceptability of the protocol. Specifically, the coaching intervention will include two parts: 1) initial coaching session with one of the study PIs, Dr. Kathryn Pollak; and 2) follow-up appointment with Dr. Pollak to check in on use of the intervention strategies. Providers will also complete self-report assessments prior to initiating CASCADE and upon completion of CASCADE. Clinic staff will let patients know that the clinic is participating in a research study about how to improve communication between patients and providers and provide patients of participating providers with an anonymous survey to complete following their clinic visit. The paper surveys will be given to all patients of the participating provider being seen in the clinic approximately 5 days prior to the coaching intervention session and 5 days following the intervention (e.g., second session with Dr. Pollak).

Descriptive statistics (e.g., means, standard deviations) will be used to characterize the experience of patients participating in focus groups with regard to their sexual functioning, emotional distress (i.e., symptoms of anxiety and depression), and physical functioning. Qualitative methods will also be used to analyze the focus groups.

Feasibility of CASCADE will be assessed by examining providers' accrual, attrition, and adherence. To determine acceptability, providers will be asked how useful the intervention was, whether the intervention will change their clinical practice, and whether they would recommend the program to a colleague. Simple t-tests will be used to examine changes in outcomes of interest (e.g., confidence, barriers, etc.) from pre- to post-intervention. Basic descriptive statistics (e.g., means, standard deviations) will be used to characterize patients' experiences during the interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients for Focus Groups: Patients treated at the Duke Cancer Institute will be recruited to participate. Patients who self-refer to the study will also be recruited to participate, and eligibility will be verified after completing informed consent. All participants will meet the following inclusion criteria: a) aged 18 years or older; b) able to speak and understand English; and c) diagnosis of breast, prostate, gynecologic, gastrointestinal, or brain cancer and treated at the Duke Cancer Institute. Patients participating in one of the two LGBTQ groups (i.e., LGBTQ individuals who identify as male; LGBTQ individuals who identify as female) must self-identify as gay, lesbian, bisexual, transgender, or queer.
* Providers: We will recruit a total of 8 providers from the Duke Cancer Institute, including 2 from each type of cancer that we are targeting (breast, gynecologic, colorectal, and prostate). Within each cancer site, we will recruit one physician and one physician-extender (physician assistant, nurse practitioner, or nurse) to represent the range of provider types. Eligible providers will be currently treating patients in one of the above listed disease groups at the Duke Cancer Institute.
* Patients recruited for CASCADE: Patients treated at the Duke Cancer Institute will be recruited to complete the anonymous survey. All participants will meet the following inclusion criteria: a) aged 18 years or older; b) able to speak and understand English; and c) diagnosis of breast, prostate, gynecologic, or gastrointestinal cancer and treated at the Duke Cancer Institute.

Exclusion Criteria:

* Patients for Focus Groups: Patients who meet any of the following criteria will be excluded: a) < 18 years old; b) cognitive or hearing impairment that is documented in the medical record, or c) unable to provide meaningful consent (i.e., severe cognitive impairment such that descriptions of the research are not clearly understood).
* Providers: Providers who treat cancers other than breast, gynecologic, colorectal, and prostate cancers will not be eligible to participate.
* Patients for CASCADE: Patients who meet any of the following criteria will be excluded: a) < 18 years old; b) cognitive or hearing impairment that is documented in the medical record, or c) unable to provide meaningful consent (i.e., severe cognitive impairment such that descriptions of the research are not clearly understood).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
PROMIS Sexual Function and Satisfaction v2 - brief profile (Sex-SF) | Focus group participants will complete this measure at the time of the focus group; up to 2 hours
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual Function and Satisfaction scale asks participants to provide information about their sexual functioning and satisfaction over the last 30 days. Separate versions of the measure will be used for males and females to address gender-specific differences in sexual functioning (e.g., pain and discomfort in the clitoris or labia vs. ability to maintain an erection). The male version of the questionnaire consists of 10 items while the female version of the questionnaire consists of 14 items. Items are assessed using a 5 point scale.
PROMIS four-item Anxiety Scale | Focus group participants will complete this measure at the time of the focus group; up to 2 hours
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item Anxiety Scale is a self-report measure of anxiety. The measures assesses fear (I felt fearful), anxious misery (i.e., My worries overwhelm me), and hyperarousal (i.e., I found it hard to focus on anything other than my anxiety), and arousal-related somatic symptoms (i.e., I felt uneasy) over the last seven days. Each item is rated on a 5 point scale ranging from 1 "never" to 5 "always." Items are summed and converted to standardized T-scores with higher scores indicative of more symptoms of anxiety. The PROMIS Anxiety Scale has been shown to have good internal reliability and convergent validity with other well validated measures of anxiety.
PROMIS four-item Depression Scale | Focus group participants will complete this measure at the time of the focus group; up to 2 hours
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item Depression Scale is a self-report measure of depressive symptoms. The measures assesses presence of depressed mood (i.e., I felt depressed, I felt hopeless, I felt helpless), as well as their self-view (e.g., I felt worthless) over the last seven days. Somatic symptoms of depression are not included in the measure as they frequently overlap with comorbid physical health concerns among medical populations. Each item is rated on a 5 point scale ranging from 1 "never" to 5 "always." Items are summed and converted to standardized T-scores with higher scores indicative of more depressive symptoms. The PROMIS Depression Scale has been shown to have good internal reliability and convergent validity with other well validated measures of depression.
PROMIS four-item Physical Function scale | Focus group participants will complete this measure at the time of the focus group; up to 2 hours
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item Physical Function scale is a self-report measure of physical functioning. The measure assesses self-reported capability of physical activities including instrumental activities (e.g., "Are you able to run errands and shop)" and mobility (e.g. "Are you able to go up and down stairs at a normal pace"). Each item is rated on a t point scale ranging from 1 "Unable to do" to 5 "Without any difficulty." Items are summed and converted to standardized T-scores, with higher scores are indicative of better physical functioning.
Psychosocial services use, preferences, and perceived barriers/facilitators questionnaire | Focus group participants will complete this measure at the time of the focus group; up to 2 hours
  A psychosocial services use, preferences, and perceived barriers/facilitators questionnaire will be completed by patients and partners/caregivers at each assessment. Participants will be asked to indicate (yes/no) whether they have utilized a list of available psychosocial services. Next, participants will indicate with yes/no to whether they have sought services for or would like services related a list of common concerns. Participants will complete a 10-item list of barriers to seeking services. Participants will state whether or not each has served as a barrier to seeking services. Finally, participants' preferences for various delivery methods will be assess. The final two questions are open ended and ask participants to list any other services they would be interested in pursuing that were not included on the list and to provide information about what might increase their use of services.
Change in confidence in talking with patients about sexuality from baseline to assessment 2 | Baseline and Assessment 2 (up to 1 year)
  Providers will be asked to rate their confidence in addressing patients' sexual health concerns using a 6-item measure. A sample item reads, Please rate state how confident you are that you can…"Initiate a discussion about a patient's sexual health concerns" (1= not at all confident to 5= very confident). The measure to be used in the present study has been adapted from a version used in our prior research (Pollak et al., 2007) and Baile et al., 1997.
Change in outcome expectancies from baseline to assessment 2 | Baseline and Assessment 2 (up to 1 year)
  Providers will be asked an adapted 6-item communication outcomes questionnaire (Parle et al., 1997) to assess possible outcomes of communication behaviors. A sample item reads, "Asking them about their sexual health concerns will benefit them" (1=very unlikely to 5= very likely). The measure to be used in the present study has been adapted from a version used in our prior research (Pollak et al., 2007) and Parle et al., 1997.
Change in comfort with sexual health discussions from baseline to assessment 2 | Baseline and Assessment 2 (up to 1 year)
  Providers will be asked to complete a 32-item measure of provider beliefs to assess their comfort with sexual health conversations. A sample item reads, "Providers focus on organic disease because they cannot treat the sexual health concerns" (1= strongly disagree to 5=strongly agree). The measure to be used in the present study has been adapted from a version used in our prior research (Pollak et al., 2007) and Ashworth et al., 1984.
Communication with providers | One time patient survey (15 minutes)
  Patients will be asked to complete several "yes" or "no" questions about whether their provider talked with them about exercise, smoking, sexual health, nutrition and sleep (e.g., did your provider talk to you about your sexual functioning during your clinic visit?). Patients will also be asked if they had wanted their provider to talk to them about the aforementioned areas using "yes" or "no" questions (e.g., Did you want your provider to talk to you about your sexual functioning during your clinic visit?).
NCCN distress screen | One time patient survey (15 minutes)
  The National Comprehensive Cancer Network (NCCN) Distress Thermometer and Problem List for Patients measures distress on a scale of zero to 10, 10 being the worst. The NCCN Problem list allows patients to inform their doctor if they are having concerns in areas such as practical, family, emotional, spiritual, and physical problems. This tool makes it easier for people to talk to their doctors about the these areas that may be affected by the diagnosis, symptoms, and treatment of cancer. Patients are encouraged to complete the NCCN Distress Thermometer and Problem List for Patients as part of their routine appointment preparation.
Service Utilization | One time patient survey (15 minutes)
  A psychosocial services use, preferences, and perceived barriers questionnaire will be completed by patients. Participants will be asked to indicate (yes/no) whether they have utilized a list of available psychosocial services. Next, participants will indicate with yes/no to whether they have sought services for or would like services related to a list of common concerns. Participants will complete a 10-item list of barriers to seeking services. Participants will state whether or not each has served as a barrier to seeking services. Finally, participants' preferences for various delivery methods will be assessed.
Usefulness of the intervention | Assessment 2 (up to 1 year)
  Providers will be asked how useful the intervention was on a 1 to 5 scale (1="Not at all useful" to 5="Extremely useful").
Likelihood the intervention would change clinical practice | Assessment 2 (up to 1 year)
  Providers will be asked the likelihood the intervention would change their clinical practice assessed on a 1 to 5 scale (1="Will not change at all" to 5="Will change a lot").
Likelihood providers would recommend the program to a colleague | Assessment 2 (up to 1 year)
  Providers will be asked the likelihood they would recommend the program to a colleague on a 1 to 5 scale (1="Definitely would not recommend" to 5="Definitely would recommend").

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Weinfurt, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided